CLINICAL TRIAL: NCT06994520
Title: Efficacy of Topical Cannabidiol in Patients With Eczema
Brief Title: Efficacy of Topical Cannabidiol for Eczema
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Khon Kaen University (Other)
Responsible Party: Principal Investigator, Suteeraporn Chaowattanapanit, Associate Professor, Khon Kaen University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HE671500
Record Dates: First submitted 2025-05-18; First posted 2025-05-29 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Chronic Pruritus; Eczema; Nummular Eczema; Atopic Dermatitis; Prurigo Nodularis
MeSH Terms: conditions — Eczema; Dermatitis, Atopic | interventions — Cannabidiol; Triamcinolone

STUDY DESIGN:
Intervention Model Description: Topical cannabidiol versus 0.1% TA cream
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cannabinoid (Experimental)
  Interventions: Other: Cannabidiol (CBD)
- Triamcinolone cream (Active Comparator)
  Interventions: Drug: Triamcinolone (TAC) 0.1% cream

INTERVENTIONS:
Other: Cannabidiol (CBD) — 5%CBD cream
  Arms: Cannabinoid
Drug: Triamcinolone (TAC) 0.1% cream — comparator
  Arms: Triamcinolone cream

SUMMARY:
Itching is a common symptom encountered in general medical practice. It can cause significant discomfort, disrupt sleep, and impair patients' quality of life. Chronic pruritic skin conditions such as atopic dermatitis, nummular eczema, lichen simplex chronicus, and prurigo nodularis are frequently observed. The pathogenesis of these conditions remains incompletely understood, and effective long-term treatment options are limited. Current therapies include topical corticosteroids, topical calcineurin inhibitors, oral corticosteroids, and systemic immunosuppressants. However, these treatments are often associated with adverse effects, and the diseases tend to follow a chronic, relapsing course. Therefore, the investigators aim to investigate the efficacy and safety of topical cannabis extract in patients with chronic pruritic skin conditions.

ELIGIBILITY:
Inclusion Criteria:

1. All participants must be aged 25 years or older.
2. Patients must be diagnosed with eczema, including atopic dermatitis, nummular eczema, lichen simplex chronicus, or prurigo nodularis, with pruritus persisting for more than 6 weeks.
3. Patients must be willing to refrain from using other topical products throughout the 4-week study period.
4. Patients must provide written informed consent to participate in the study.

Exclusion Criteria:

1. Patients who have taken oral steroids, immunosuppressive drugs, or received phototherapy within the past 3 months.
2. Patients with chronic kidney disease, liver cirrhosis, cancer, or thyroid disease.
3. Pregnant or breastfeeding women, or women planning to become pregnant.
4. Patients who develop erythematous itchy rash in response to an open patch test using cannabis extract products.
5. Patients with a known allergy to cannabis-derived products, which may result from other ingredients and/or solvents used in the extraction process.
6. Patients with severe or unstable cardio-pulmonary diseases (e.g., angina, peripheral vascular disease, cerebrovascular disease, or arrhythmia), or those at risk of cardiovascular disease.
7. Patients with a history of psychosis, current active mood disorder, or anxiety disorder.
8. Patients who are addicted to substances, including nicotine, or are heavy alcohol users.
9. Patients using other medications, particularly opioids or sedatives such as benzodiazepines.
10. Patients taking medications known to potentially interact with cannabis extracts, such as warfarin, fluoroquinolones, or dihydropyridine calcium channel blockers.

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Disease severity | 4 weeks
  Disease severity was evaluated using a composite scoring system that assessed four clinical signs-erythema, induration, scaling, and scratching-along with the extent of area involvement. Each sign was graded on a 4-point scale: 0 = none, 1 = mild, 2 = moderate, and 3 = severe. The extent of area involvement was classified into six categories based on the percentage of body surface area affected: 1 = less than 10%; 2 = 10-<30%; 3 = 30-<50%; 4 = 50-<70%; 5 = 70-<90%; 6 = 90-100%.
  The overall severity score was obtained by summing the individual scores for erythema, induration, scaling, and dryness for each affected area and then multiplying this sum by the corresponding area involvement score. Higher total scores indicated greater disease severity.
Changing of erythema | 4 weeks
  Erythema was graded on a scale from 0 to 3, with 0 indicating no redness, 1 mild, 2 moderate, and 3 severe redness.
Changing of induration | 4 weeks
  Induration was graded on a scale from 0 to 3, with 0 indicating no induration, 1 mild, 2 moderate, and 3 severe skin thickening.
Changing of scaling | 4 weeks
  Scaling (flaking of the skin) was graded on a scale from 0 to 3, with 0 indicating none, 1 mild, 2 moderate, and 3 severe.
Changing of scratching | 4 weeks
  Excoriation (scratching marks) was graded on a scale from 0 to 3, with 0 indicating no excoriation, 1 mild, 2 moderate, and 3 severe excoriation.
Itching severity | 4 weeks
  Itching severity was assessed using an 11-point numeric rating scale (NRS). The NRS-11 evaluates average intensity of pruritus ranging from 0 (no itch) to 10 (worst imaginable itch). Scores were classified into three groups as follows: 0-3 = mild, 4-7 = moderate, and 8-10 = severe.

SECONDARY OUTCOMES:
Adverse events | 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Khon Kaen University, Khon Kaen, Changwat Khon Kaen, Thailand